CLINICAL TRIAL: NCT00050986
Title: Phase I/II Evaluation Temozolomide and Farnesyl Transferase Inhibitor ZARNESTRA (R115777) for the Treatment of Recurrent and Progressive Glioblastoma Multiforme
Brief Title: Phase I/II Evaluation of Temozolomide and ZARNESTRA (R115777) for Recurrent and Progressive Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-126
Record Dates: First submitted 2002-12-31; First posted 2003-01-03 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Glioblastoma Multiforme
Keywords: Brain Neoplasms; CNS Diseases; Glioblastoma Multiforme; Temozolomide; Temodar; R115777; Zarnestra
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Central Nervous System Diseases | interventions — Temozolomide; tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide and R115777 (Experimental)
  Interventions: Drug: Temozolomide; Drug: R115777

INTERVENTIONS:
Drug: Temozolomide — Starting Dose Level: 100 mg/m^2 taken by mouth once daily for 7 days, followed by 7 days rest and another 7-day dosing period and 7-day rest period.
  Other Names: Temodar
Drug: R115777 — Starting Dose Level: 400 mg taken by mouth for 7 consecutive days every other week on alternating weeks (days 8-14 and 22-28) every 4 weeks.
  Other Names: Zarnestra

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of the new drug ZARNESTRA (R115777) and temozolomide that can be given to patients with brain tumors (glioblastoma multiforme, GBM). The second goal is to learn if these drugs given in combination can shrink or slow the growth of brain tumors. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Temozolomide works by killing cancer cells. R115777 is a new drug that may slow down the growth of cancer cells. Used in combination, the two drugs may control the growth of brain tumors.

Before treatment starts, patients will have a complete exam, including measurement of height and weight. Blood tests (less than 2 tablespoons of blood) will be performed. A MRI scan will be done. Women who are able have children must have a negative blood pregnancy test.

Temozolomide and R115777 will both be taken by mouth. Participants in this study will take temozolomide once a day for 7 days every other week (Days 1-7 and 15-21). This will be repeated every 28 days (1 course). Patients must not eat for 1 hour before and after taking the drug; drinking water is allowed. All treatment may be given on an outpatient basis.

During the alternate weeks (Days 8-14 and 22-28), participants will take R115777 tablets by mouth in the morning and evening with food. At the beginning of the study, groups of 3 participants each will take increasing doses of both R115777 and temozolomide until the highest safe dose of each drug, when given in combination, is found. Participants entering the study after the highest safe dose is found will receive that dosage.

If tumors do not grow and serious side effects do not occur, participants may keep on taking temozolomide and R115777 for up to 2 year. If your physician thinks it is advisable, treatment may continue with R115777 alone after that time. In this case, routine blood tests for counts, liver and kidney function (less than 2 tablespoons) will be repeated every 4 weeks and MRI scans, physical, and neurological exams will be done every 8 weeks. Participants may not receive any other treatment for cancer (including surgery) while taking part in this study.

Participants will come to the clinic to have a complete physical and neurological exam and blood tests (less than 2 tablespoons of blood) before each course. Blood tests will be repeated once a week for the first 2 courses of treatment and then on Days 14 and 28 of each later course. A MRI scan will be done before the odd-numbered (3, 5, 7, etc.) courses of treatment or at any time clinically indicated.

At the end of the study, participants will have another complete physical exam. Blood tests (less than 2 tablespoons of blood) will be performed. A MRI scan will be done.

This is an investigational study. Temozolomide is approved by the FDA for the treatment of some brain tumors and is commercially available. R115777 is approved for research use only in the treatment of brain tumors. The use of these two drugs together is experimental.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven supratentorial glioblastoma multiforme (GBM).
2. Patients must have shown unequivocal evidence for tumor recurrence or progression by MRI scan after radiation therapy. The scan done prior to study entry documenting progression will be reviewed by the primary investigator to document tumor volume changes to provide a gross assessment of growth rate.
3. Patients may have had: a) no prior chemotherapy, b) 1 prior adjuvant chemotherapy, c) 1 prior adjuvant chemotherapy followed by 1 regimen for recurrent disease, or d) 1 or 2 prior chemotherapy regimens for recurrent or progressive tumor.
4. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of this hospital.
5. Patients must have shown unequivocal evidence for tumor progression by MRI or CT scan. A scan should be performed within 14 days prior to registration and on a steroid dose that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement.
6. Pts with recent resection of recurrent or progressive tumor will be eligible if all of the following conditions apply: Pt has recovered from the effects of surgery; Residual disease after resection of recurrent tumor is not mandated for eligibility. To assess the extent of residual disease post-operatively, a CT/MRI should be done no later than 96 hours post-operatively or at least 4 weeks post-operatively, and within 14 days before registration. If steroid dose increased between the day of imaging and registration, a new baseline scan is required after stable steroids for 5 days.
7. Patients must have a Karnofsky performance status of >/= 60
8. Patients must have recovered from the toxic effects of prior therapy: 4 weeks from prior cytotoxic therapy and/or at least two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
9. Patients must have adequate bone marrow function (ANC>/= 1,500/mm(3) and platelet count of >/= 100,000/mm(3)), adequate liver function (SGPT and SGOT </= 2.5 times normal, bilirubin </= 2 mg%), and adequate renal function (BUN and creatinine <1.5 times institutional normal) prior to starting therapy.
10. ZARNESTRA may interfere with coumadin dosing and patients who are taking this combination will require more frequent monitoring of their PT, PTT and INR.
11. Patient has no risk factors for HIV or is serologically negative.

Exclusion Criteria:

1. Patients must not be taking primidone, carbamazepine, phenobarbital or phenytoin anticonvulsants. Patients changing from these anticonvulsants to others that are allowed must be off the drugs listed above for at least 1 week.
2. Patients must not be taking cimetidine, erythromycin azole antifungals, paclitaxel, tacrolimus or cyclosporine.
3. Patients must not have uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, myocardial infarction within the previous six months, or serious uncontrolled cardiac arrhythmia.
4. Because of the concerns of potentially harmful interactions of ZARNESTRA and other medications taken by patients who are HIV positive or have AIDS related diseases, patients who are HIV positive will not be eligible for entry into this study. Only patients with suspected HIV will be tested and if positive, will be ineligible.
5. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) are ineligible unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
6. Patients must not have: a) active infection b) disease that will obscure toxicity or dangerously alter drug metabolism c) serious intercurrent medical illness. d) prior recurrence with either Temozolomide or a farnesyl transferase inhibitor.
7. Patients must not be pregnant and must practice adequate contraception

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2002-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Gilbert, Principal Investigator — MDAnderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 55 participants recruited in between 12/30/2002 and 11/30/2005, all at M. D. Anderson Cancer Center.
Pre-assignment Details: 5 patients were not evaluated for response because of the following: 1 early, non-treatment related death; 3 withdrew consent; 1 discontinued for intercurrent illness (pneumonia).
Period: Overall Study
Arm/Group | Temozolomide and R115777
Started | 55
Completed | 53 (Two participants had withdrawn consents before the study treatment was initiated.)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide and R115777
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 52 [21 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Maximal Tolerating Dose (MTD for Phase I)
Description: Phase I Dose limiting toxicity evaluation at end of first cycle based on blood tests every two weeks and participants' subjective and objective symptoms.
  Start Dose Level 100 mg/m² Temozolomide once daily + 400 mg ZARNESTRA twice daily; Dose Level 1 100 mg/m² Temozolomide once daily + 500 mg ZARNESTRA twice daily; Dose Level 2 150 mg/m² Temozolomide once daily + 500 mg ZARNESTRA twice daily; Dose Level 3 150 mg/m² Temozolomide once daily + 600 mg ZARNESTRA twice daily; Dose Level 4 150 mg/m² Temozolomide once daily + 800 mg ZARNESTRA twice daily
Time Frame: End of first cycle (4 weeks) evaluation
Population: As treated.
Measure: Number; unit: participants
Arm/Group | Temozolomide and R115777
Number analyzed (Participants) | 15
participants
  Dose Level 1 | 3
  Dose Level 2 | 3
  Dose Level 3 | 6
  Dose Level 4 | 3

2. Secondary Outcome: Progression-free Survival (Phase II)
Description: Efficacy measured by 6 month progression-free survival assessment.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years, 11 months
Description: Including all serious adverse events regardless of attribution. Including all grade 3 or higher adverse events regardless of attribution.
Arm/Group | Temozolomide and R115777
Serious Adverse Events (participants affected / at risk) | 24/53
Other Adverse Events (participants affected / at risk) | 47/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide and R115777 (N=53)
Thrombosis/embolism (Vascular disorders) | 4 (4) — Pulmonary Embolism and deep vein thrombosis
Seizure (Nervous system disorders) | 3 (3)
Death (Nervous system disorders) | 2 (2) — Due to tumor progression. Not related to the study drugs
Neutrophils (Blood and lymphatic system disorders) | 3 (3)
confusion (Nervous system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Herpes Zoster (Infections and infestations) | 2 (2)
Depressed level of consiousness (Nervous system disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 2 (2)
hypophasphatemia (Metabolism and nutrition disorders) | 1 (1)
Pyramidal Tract Dysfunction (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection (Infections and infestations) | 5 (5)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
CNS Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Amyliase, Lipase, Pancreatitis (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide and R115777 (N=53)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
ALT (Metabolism and nutrition disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 5 (6)
Anorexia (Gastrointestinal disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4)
decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 7 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (11)
Neutrophils (Blood and lymphatic system disorders) | 21 (76)
Hearing (Ear and labyrinth disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5)
Hypotension (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphocytopenia (Blood and lymphatic system disorders) | 40 (210)
Mental Status (Nervous system disorders) | 3 (3)
Motor (Nervous system disorders) | 6 (6)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain (General disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 1 (1)
Personality/behavioral (Nervous system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (30)
Pneumonits (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Seizures (Nervous system disorders) | 4 (4)
Speech impairment (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis (Blood and lymphatic system disorders) | 3 (3)
Weight gain (General disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes